CLINICAL TRIAL: NCT02109263
Title: Breastfeeding Versus Saccharose for Prevention of the Procedural Pain in the Newborn
Brief Title: Prevention of the Procedural Pain in the Newborn
Acronym: ACTISUCROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RB 12.143
Record Dates: First submitted 2013-07-10; First posted 2014-04-09 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2015-04

CONDITIONS: Prevention of the Procedural Pain in the Newborn
Keywords: Breast-feeding; Saccharose; Breast-feeding newborn; cortical pain responses; near infrared spectroscopy (NIRS); Salivary rate cortisol; heel lance
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saccharose (Experimental): 20% saccharose
  Interventions: Procedure: saccharose versus breast-feeding
- breast-feeding (Placebo Comparator): breast-feeding
  Interventions: Procedure: saccharose versus breast-feeding

INTERVENTIONS:
Procedure: saccharose versus breast-feeding — saccharose versus breast-feeding

SUMMARY:
The aim of this study is to compare the impact of two non-medicinal strategies: the breast-feeding and saccharose to measure effects in cerebral cortex during pain using near infrared spectroscopy (NIRS)

DETAILED DESCRIPTION:
Many studies of non-medicinal treatments(saccharose and breast-feeding)show a decrease of expression of pain in newborn. However Slater and al questioned these practices due to the absence of modification of the cerebral answer measured by evoked potential.

ELIGIBILITY:
Inclusion Criteria:

* Gestationnel age included between 37 and 42 weeks
* Born in the CHRU of Brest
* Breast-Fed
* Score of Apgar upper to 7
* No pathology malformative
* Absence of known chromosomal abnormality
* Consent of parents

Exclusion Criteria:

* Maternal drug use
* Morphinic treatment
* Barbiturate treatment
* Benzodiazépine treatment

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Increase of the total concentration of haemoglobin | Measure two minutes before painful gesture, at the moment of painful gesture and 2 minutes after painful gesture. The newborn will be followed for the duration of hospital stay, an expected average of 30 to 60 minutes
  Increase of the total concentration of haemoglobin (delta HbT) measured by the spectrometer during the intravenous injection.

SECONDARY OUTCOMES:
Dosage of rate salivary cortisol | before and after painful gesture
  Salivary cortisol sampling

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel ROUE, Principal Investigator — Pole de la femme, de la Mère et de l'Enfant, CHRU de Brest
Locations (1):
- Centre hospitalier universitaire, Brest, France

REFERENCES:
- [Result] Rioualen S, Durier V, Herve D, Misery L, Sizun J, Roue JM. Cortical Pain Response of Newborn Infants to Venepuncture: A Randomized Controlled Trial Comparing Analgesic Effects of Sucrose Versus Breastfeeding. Clin J Pain. 2018 Jul;34(7):650-656. doi: 10.1097/AJP.0000000000000581. PMID 29298184